CLINICAL TRIAL: NCT00181701
Title: A Phase II Trial of Intraperitoneal Paclitaxel and Carboplatin Therapy in the Treatment of Women With Newly Diagnosed, Optimally Cytoreduced Carcinoma of Mullerian Origin
Brief Title: Intraperitoneal Paclitaxel and Carboplatin in the Treatment of Women With Carcinoma of Mullerian Origin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Richard Thomas Penson, Clinical Director Medical Gynecologic Oncology, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-100
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Ovarian Carcinoma
Keywords: Ovarian cancer; Epithelial carcinoma of mullerian origin; Intraperitoneal paclitaxel; Intraperitoneal carboplatin; Primary peritoneal carcinoma; Tubal carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
The main purpose of this study is to determine the safety and tolerability of giving both paclitaxel and carboplatin in the abdominal cavity by looking at what effects (good and bad) this route of administration has on patients with ovarian cancer. Standard chemotherapy drugs are administered intravenously but a number of trials have shown that injecting drugs into the abdominal cavity, or intraperitoneally, have shown promising results.

DETAILED DESCRIPTION:
Patients will have an intraperitoneal port placed at the time of their initial surgery or at a second procedure prior to cycle 2 of chemotherapy.

Patients will receive a total of 6 cycles of therapy as an outpatient. They will have 1 cycle of paclitaxel/carboplatin intravenously followed by 5 cycles of paclitaxel/carboplatin intraperitoneally. Chemotherapy treatment is given on days 1, 8, and 15 of each cycle. Each cycle is 21 days long.

To help reduce the chance of an allergic reaction, patients will also take decadron tablets orally before paclitaxel administration.

About 1 liter of standard salt solution will be injected through a catheter into the abdominal cavity with each treatment to help distribute the drugs throughout the abdominal cavity.

"Second-look" surgery (laparoscopy or laparotomy) will be performed 3-8 weeks after the last chemotherapy course (cycle 6) if the patient is in complete clinical remission. This surgery is done to see how effective the chemotherapy was.

Tests and procedures will be done throughout the treatment to see how the cancer is responding and to monitor for safety purposes. These tests and procedures include routine history and physical exam, neurological exam, and routine blood tests. As part of this study we will also be checking the amount of paclitaxel and carboplatin in the blood.

Participation in this study will last approximately 6 months as long as the treatment is well tolerated, there are no serious side effects and the disease has not progressed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial carcinoma of mullerian origin. Specifically, ovarian, primary peritoneal and tubal carcinoma
* Stage II or III disease
* Patient must have undergone surgical staging and debulking with optimal cytoreduction
* Able and willing to undergo a second look staging laparotomy
* 18 years of age or older
* Adequate bone marrow function with an Absolute Neutrophil Count (ANC) > 2,500 and platelets > 100,000/mm3
* ECOG performance status less than or equal to 2

Exclusion Criteria:

* Disease outside the abdominal cavity
* Stage IV disease, including abdominal wall, visceral and/or pleural involvement
* Previous chemotherapy for ovarian cancer
* Suboptimal cytoreduction
* Creatinine > 1.5 mg/dl
* History of recent Myocardial Infarction or congestive heart failure within 6 months of surgery
* SGOT > 2x Upper Limit of Normal (ULN), bilirubin > 1.5 x ULN
* Colostomy or ileostomy
* Concurrent invasive malignancy
* Known hypersensitivity to E. coli derived products
* Active psychiatric or mental illness precluding informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of carboplatin and paclitaxel administered intraperitoneally

SECONDARY OUTCOMES:
To determine the efficacy of this regimen as defined by surgical response rate

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Penson, MD, Principal Investigator — Massachusetts General Hospital